CLINICAL TRIAL: NCT04272398
Title: An Investigation of the Effects of Dynamic Elastomeric Fabric Orthoses Used for Lower Body and Pelvis in Children With Cerebral Palsy on Balance, Gait Parameters, and Pelvic Symmetry
Brief Title: Effects of Using Dynamic Elastomeric Fabric Orthoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Sabiha BEZGİN, Physical Therapist, Kırıkkale University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: Kirikkale U
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy; Movement Disorders; Neurologic Disorder
Keywords: cerebral palsy; dynamic orthoses; gait analysis; movement; neoprene; rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Movement Disorders; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Used dynamic elastomeric fabric orthoses with physiotherapy and rehabilitation program
  Interventions: Other: dynamic elastomeric fabric orthoses
- Control (Experimental): Only physiotherapy and rehabilitation program
  Interventions: Other: dynamic elastomeric fabric orthoses

INTERVENTIONS:
Other: dynamic elastomeric fabric orthoses — Wore dynamic elastomeric fabric orthoses with a focus on the lower body and pelvis in addition to the physiotherapy and rehabilitation sessions. The frequency of the use of the orthosis was planned to extend through the week and they had the orthosis during their active hours during the day about 8 hours a day.

SUMMARY:
Purpose: The aim of this study was to investigate the effects of dynamic elastomeric fabric orthoses (DEFOs) used for lower trunk and pelvis on balance, gait parameters, and pelvis symmetry in children with cerebral palsy.

Materials and Methods: Twenty-two children (7 girls, 15 boys) in an age range of 4-10 years, with spastic type cerebral palsy, and at gross motor function classification system levels 1 or 2 were included in the study. Children who met the inclusion criteria were randomly divided into two groups. Ten children were included in the control group (Group I) and 12 children were included in the orthosis group (Group II). Both groups received a physiotherapy and rehabilitation program twice a week for 8 weeks in accordance with neurodevelopmental treatment approaches. Children in Group II were treated with DEFOs in lower body and pelvis in addition to physiotherapy and rehabilitation sessions. The use frequency of the orthosis was extended over the course of the week during which they were active for 8 hours a day. After the demographic data of the children were recorded, the Pediatric Balance Scale and the Timed Up and Go Test were used for balance assessment. Gait parameters and kinematic values of the pelvis were evaluated using the BTS G-Walk®, a wireless mini digital gait analysis system.

DETAILED DESCRIPTION:
All groups received a physiotherapy and rehabilitation program two sessions per week, for 45 minutes, for a total of 8 weeks. The program was administered by a physiotherapist and prepared in accordance with neurodevelopmental treatment approaches. At other times, families continued to practice the exercises. An appropriate treatment plan was developed according to the needs and characteristics of each participant. Ensuring proper posture in different positions, increasing body awareness, and facilitating trunk extension were included in the treatment plan. For the development of postural control in standing and walking without support, weight transfer studies on the affected and less affected sides with trunk elongation were emphasized. Step up/down exercises were performed on both the affected and less affected sides. Supported by appropriate hand gripping, two-feet forward jumping, one-foot forward jumping, and weight transfer on one leg exercises were performed. Providing sensory inputs during all exercises was given importance. Exercises were conducted particularly to strengthen the antagonists of the spastic muscles. Stretching exercises were carried out in functional positions with active participation of the child as much as possible. The home program was shown to the family in detail in parallel with the physiotherapist's practices and the program was revised regularly. While Group I continued physiotherapy and rehabilitation sessions, the children in Group II wore DEFOs with a focus on the lower body and pelvis in addition to the physiotherapy and rehabilitation sessions. The frequency of the use of the orthosis was planned to extend through the week and they had the orthosis during their active hours during the day about 8 hours a day. In order to reduce the loosening of the fabric caused by extensive use, it was recommended that the orthosis be removed and reworn at two-hour intervals. The children wore the DEFOs for 8 weeks with this frequency. The frequency of use was monitored using a chart. Children were evaluated at the beginning of the study and after 8 weeks. An assessment environment was created for each child when they felt energetic and well. In order to prevent fatigue, short breaks were given. All evaluations were performed in the same environment in standardized conditions and without orthosis. Gait analysis was performed with bare feet.

ELIGIBILITY:
Inclusion Criteria:

* Both the child and the family need to volunteer to participate in the study, diagnosis of spastic type CP with bilateral or unilateral involvement,
* being at level 1 or 2 based on the Gross Motor Function Classification System (GMFCS) and
* being in an age range of 4-10 years.

Exclusion Criteria:

* who had received botulinum toxin/surgery at the lower extremity and/or pelvis in the previous six months and those who were going to receive this treatment during the study were excluded from the study.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Balance | 8 weeks
  Second with Time and go test
Walking speed | 8 weeks
  (meter/second)
Stance phase | 8 weeks
  its percentage within gait cycle
Swing phase | 8 weeks
  its percentage within gait cycle
Symmetry Index of Pelvic Movements | 8 weeks
  percentage

SECONDARY OUTCOMES:
Step length | 8 weeks
  its percentage within two-step length
Single support phase | 8 weeks
  its percentage within two-step length

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Bezgin, PhD, Principal Investigator — Kırıkkale University
Locations (1):
- Kırıkkale University, Kırıkkale, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bezgin S, Novak I, Cobanoglu G, Elbasan B. Effects of dynamic elastomeric fabric orthoses in children with cerebral palsy: A single-blind randomized controlled trial. Prosthet Orthot Int. 2025 Apr 1;49(2):220-227. doi: 10.1097/PXR.0000000000000425. Epub 2024 Dec 24. PMID 39721059